CLINICAL TRIAL: NCT00115752
Title: Genetic Basis For Variation In NSAID Analgesia In A Clinical Model Of Acute Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050176; 05-NR-0176
Record Dates: First submitted 2005-06-23; First posted 2005-06-24 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2006-10-04

CONDITIONS: Pain
Keywords: Single Nucleotide Polymorphism; Analgesic Efficacy; Oral Surgery Model; Cyclooxygenase Inhibitor; Gene Expression Profile; Wisdom Teeth; Third Molar Extraction
MeSH Terms: conditions — Pain | interventions — valdecoxib; Cyclooxygenase Inhibitors

INTERVENTIONS:
Drug: Valdecoxib
Drug: COX Inhibitor

SUMMARY:
This study will evaluate how genetic makeup contributes to the variation in people regarding their sensitivity to and experience of pain. Scientists believe that differences in information found in genes may explain why an analgesic drug, that is, one that treats pain, works effectively for some people but not for others. The study will explore pain that is acute (fast and short period). Knowledge gained from this ongoing study may permit development of an individualized analgesic drug prescription.

Patients ages 16 to 35 who are in good health and have been referred for removal of impacted wisdom teeth; who are not allergic to aspirin or other nonsteroidal anti-inflammatory drugs (known as NSAIDs), sulfites, or certain anesthetics; who are not pregnant or nursing; and who are willing to have a biopsy before and after dental surgery are eligible for this study.

Patients will come to the clinic for one test visit and one treatment visit. During the first visit, a questionnaire will evaluate patients' psychological state, including mood and depression. There will be a clinical examination of their wisdom teeth. A blood sample of 10 milliliters (about 0.4 ounces) will be collected from the forearm to provide DNA material containing genes stored in cells. The primary genetic analysis will be done at NIH, although the DNA collected might also be sent to a laboratory outside NIH. DNA samples will be coded so that names of patients cannot be traced.

During the second visit, two of the patients' lower wisdom teeth will be removed. Patients will be given a local anesthetic in the mouth and a sedative given through a vein in the arm. While the mouth is numb, a small piece of tissue will be removed from inside the cheek, near the wisdom tooth. It is the first biopsy. After the two wisdom teeth are removed, a small piece of tubing will be placed into both sides of the mouth where the teeth were removed. Every 20 minutes, for the next 3 hours, the researchers will collect inflammatory fluid from the tubing, to measure the chemicals thought to cause pain and swelling. Also every 20 minutes, patients will rate the pain they feel by answering questions. If there is pain before 3 hours following surgery, they will receive a dose of fentanyl to relieve moderate to severe pain. A second biopsy will occur 3 hours after surgery, to measure changes in chemicals produced in response to surgery. Immediately afterward, patients will receive 30 mg of ketorolac (Toradol) whether or not pain is felt. They will answer questionnaires about pain for 3 hours after receiving the drug, to rate how well it works. They will stay at the clinic up to 6 hours after the surgery. If pain is not relieved with ketorolac, patients will receive a one-time dose of tramadol, a pain medication for moderate to severe pain. After the study procedures are completed, patients will receive pain medication for pain after surgery.

Patients will be monitored closely, because all drugs have side effects. Ketorolac is a nonsteroidal anti-inflammatory drug, one that may cause gastrointestinal upset. Fentanyl is a powerful narcotic drug that is safe at the dosage used in this study, but stomach upset, dizziness, and breathing trouble may occur. Also, risks from the biopsy include discomfort from injecting the numbing medicine, infection, and bleeding. There may be discomfort from the sedative injected into the vein, and there may be bruising.

Benefits from participating are having wisdom teeth removed at no cost as well as close monitoring before and after surgery. There are no plans to give patients the results of genetic tests or questionnaires. Years of research may be needed before such information has the chance to become meaningful.

DETAILED DESCRIPTION:
The proposed clinical trial will evaluate the role of genetic factors including single nucleotide polymorphisms from cyclooxygenase (COX) - 2 gene on acute pain after tissue injury and the analgesic effect of a COX inhibitor. Patients will be healthy volunteers scheduled for the surgical removal of impacted third molars. Genotyping will be performed before surgery and patients stratified to treatment with a COX inhibitor in this protocol or to other protocols examining different polymorphisms.

Under local anesthesia, 2 mandibular third molars will be removed. Microdialysis sampling in the extraction socket will be performed with pre- and post-surgical biopsies. Patients will receive a COX inhibitor as an analgesic drug for the post-operative pain. Outcomes evaluated will include clinical pain response, gene expression profile using microarray and quantitation of related proteins after oral surgery and the interaction of these factors with analgesia by a COX inhibitor. By studying these responses in patient samples for each genotype (non-variant homozygote, heterozygote and variant homozygote) from the COX-2 gene, we will attempt to replicate and extend previous findings on the role of genetic factors in the inflammatory process, clinical pain and variation in response to analgesic drugs.

ELIGIBILITY:
* INCLUSION CRITERIA

Male or female volunteers referred for third molar extraction willing to undergo 2 visits: 1 test and blood withdrawal visit and 1 surgical appointment

Between the ages of 16 to 35 years (based upon eruption patterns and age-related complications associated with surgical extraction of third molars)

In general good health- American Society of Anesthesiologists (ASA) status I or II (healthy subjects based upon criteria for safe administration of out-patient conscious sedation)

Willing to undergo observation period for up to 6 hours postoperatively (3 hours post-surgery and 3 hours post-medication)

Ability to complete a 100 mm VAS and a category scale every 20 minutes for the observation period (6 hours)

Willing to have a microdialysis probe placed beneath the surgical flap during the 3 hours post-surgery and 3 hours post-medication

Willing to have a preoperative and postoperative biopsy at 3 hours after the surgery

Must have two lower partial (rating = 3) or fully impacted (rating = 4) wisdom teeth (mandibular third molars)

As assessed at the screening visit, the sum of the mandibular third molar surgical difficulty ratings must be between 6 to 8 in order to evaluate subjects experiencing similar pain levels

As assessed at the screening visit, subjects must have specific ethnic background of interest to minimize the ethnic effect on pain sensitivity, genotype frequency and haplotype patterns.

As assessed at the genotyping, subjects must have specific genotype of interest

EXCLUSION CRITERIA

Patients who are allergic to aspirin, NSAIDs, sulfites, or amide anesthetics

Patients who have had asthma, or hives

Patients who are pregnant or nursing

Patients with history of peptic ulcers and/or GI bleeding

Ages: 7 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 96
Dates: Start 2005-06-20; Study Completion 2006-10-04

PRIMARY OUTCOMES:
Clinical pain response.

SECONDARY OUTCOMES:
Gene expression profiles using microarray and quantitation of related proteins after oral surgery and the interaction of these factors with analesia by a COX inhibitor.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Nursing Research (NINR), Bethesda, Maryland, United States

REFERENCES:
- [Background] Gordon SM, Brahim JS, Dubner R, McCullagh LM, Sang C, Dionne RA. Attenuation of pain in a randomized trial by suppression of peripheral nociceptive activity in the immediate postoperative period. Anesth Analg. 2002 Nov;95(5):1351-7, table of contents. doi: 10.1097/00000539-200211000-00047. PMID 12401625